CLINICAL TRIAL: NCT00369304
Title: A Randomized, Open Label, 2-Period Crossover Study to Determine the Pharmacokinetics of the Potential Drug Interaction Between CYP2C9 Inhibitor and Substrate.
Brief Title: Study Evaluating the Pharmacokinetics of the Potential Drug Interaction Between CYP2C9 Inhibitor and Substrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3189A1-103
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Subjects
Keywords: Health
MeSH Terms: interventions — Drug Interactions

INTERVENTIONS:
Drug: pharmacokinetic (how the body absorbs and eliminates) interaction

SUMMARY:
This is an open-label, randomized, 2-period crossover, inpatient study to be performed in healthy subjects. The study will consist of 2 treatment periods: There will be 2 parallel cohorts of 12 subjects each who will be enrolled to receive single doses of tolbutamide or AGG-523 plus tolbutamide in periods 1 and 2 in a crossover design. Doses of test article will be administered after an overnight fast of at least 10 hours.

ELIGIBILITY:
1. Men and women, aged 18 to 50 years. Women of non-childbearing potential may be included.
2. Body mass index in the range of 18 to 30 kg/meter squared and body weight equal to or greater than 50 kg.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12 lead electrocardiogram (graphic trace of the pattern of your heart beat).
4. Non-smoker or smoker of fewer than 10 cigarettes (half a pack) per day as determined by history. Must abstain from smoking during inpatient stay.
5. Have a high probability for compliance with and completion of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of a single oral dose of AGG-523 on the pharmacokinetic profile of a single oral dose of tolbutamide in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer